CLINICAL TRIAL: NCT01633671
Title: NT-proBNP: a Useful Tool for the Detection of Acute Pulmonary Artery Embolism in Post-surgical Patients
Brief Title: NT-proBNP as a Tool for the Detection of Acute Pulmonary Artery Embolism (APE)
Status: Completed | Type: Observational
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Claus-Martin Muth, Claus-Martin Muth, MD, PhD - Head of the Department of Emergency Medicine, University of Ulm
Other Study IDs: ana-ulm-ntprobnp-288/11
Record Dates: First submitted 2012-06-28; First posted 2012-07-04 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Pulmonary Embolism; Pulmonary Embolism Without Mention of Acute Cor Pulmonale
Keywords: Misadventures to Patients During Surgical and Medical Care; Pulmonary Embolism Without Acute Cor Pulmonale; Pulmonary Embolism Without Mention of Acute Cor Pulmonale
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suspected APE: Post-surgical patients with clinically suspected acute pulmonary embolism

SUMMARY:
In patients with suspected APE (Acute Pulmonary Embolism) referred to the intensive care unit (ICU)after major surgery, serum NT-proBNP (N-terminal proBNP), Troponin-I and D-dimers were measured according to the standard hospital protocol. To definitively confirm or exclude APE, all patients underwent an angiographic CT-scan of the thorax.

DETAILED DESCRIPTION:
In patients with suspected APE referred to the intensive care unit after major surgery, serum NT-proBNP, Troponin-I and D-dimers were measured according to the standard hospital protocol. Blood samples were obtained within one hour after the onset of clinical symptoms.

Definitive confirmation or exclusion of APE was performed with an angiographic CT-scan of the thorax.

ELIGIBILITY:
Inclusion Criteria:

all patients referred to the ICU with suspected APE

Exclusion Criteria:

none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients after major surgery referred to the anesthesiologic ICU due to suspected acute pulmonary embolism.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2008-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Acute pulmonary embolism: CT-proof yes vs. no | 1 hour after onset of clinical symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Claus M Muth, MD, Study Chair — Dept. of Anesthesiology, Div. of Emergency medicine, University hospital Ulm, 89075 Ulm, Germany; Bernd E Winkler, MD, Principal Investigator — Dept. of Anesthesiology, University hospital Ulm, 89075 Ulm, Germany
Locations (1):
- University of Ulm, Michelsberg anaesthesiologic ICU, Ulm, Baden-Wurttemberg, Germany